CLINICAL TRIAL: NCT04935086
Title: Risk Factors for Predictors of Major Adverse Cardiovascular Events After Coronary Artery Bypass Using Radial Artery Grafts
Brief Title: Risk Factors for Predictors of MACEs After RA-CABG
Status: Completed | Type: Observational
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Qiang Zhao,MD, Professor and Director, Department of Cardiovascular Surgery, Vice President, Ruijin Hospital, Ruijin Hospital
Other Study IDs: KY-2020388
Record Dates: First submitted 2021-06-03; First posted 2021-06-22 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Coronary Artery Disease
Keywords: Risk Factors; CABG; Radial Artery; MACE
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- MACE Group: MACE Group includes the patients suffered from any component of MACE after RA-CABG until the latest follow-up.
- Non-MACE Group: Non-MACE Group includes the patients freed from any component of MACE after RA-CABG until the latest follow-up.

SUMMARY:
As the secondary choice of artery grafts, radial artery is more and more used to achieve multiple arterial revascularization in CABG. Risk factors for predictors of major cardiovascular adverse events (MACE) after CABG using radial-artery grafts (RA-CABG), however, remain uncertain. This case-control study aims to identify the baseline predictors of MACE after RA-CABG.

We will collect the baseline characteristics and perioperative data of patients underwent RA-CABG from Jan. 2009 to Dec. 2019 in our single center. By reviewing the latest follow-up records, we will examine the correlation between the baseline characteristics and clinical outcomes (MACEs), then identify the independent risk factors for predictors of MACEs after RA-CABG.

ELIGIBILITY:
Inclusion Criteria:

* Underwent CABG using at least a radial artery grafts from Jan.2009 to Dec.2019. with or without cardiopulmonary bypass , with or without concomitant procedure
* Aged 18 and above at procedure
* With any gender

Exclusion Criteria:

* With unavailable medical records

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 18-year and above underwent RA-CABG from Jan. 2009 to Dec.2019 in one single center.
Sampling Method: Probability Sample
Enrollment: 370 (Actual)
Dates: Start 2021-06-30 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
7-day MACE-4 | 7 days post-CABG
  a composite of all-cause death, myocardial infraction, stroke and repeat revascularization
30-day MACE-4 | 30 days post-CABG
  a composite of all-cause death, myocardial infraction, stroke and repeat revascularization
1-year MACE-4 | 1 year post-CABG
  a composite of all-cause death, myocardial infraction, stroke and repeat revascularization
3-year MACE-4 | 3 years post-CABG
  a composite of all-cause death, myocardial infraction, stroke and repeat revascularization

SECONDARY OUTCOMES:
MACE-3 | 7 days, 30 days, 1 year, and 3 years post-CABG
  a composite of CV-death, myocardial infraction and stroke
All-cause death | 7 days, 30 days, 1 year, and 3 years post-CABG
  Death from any cause
CV-death | 7 days, 30 days, 1 year, and 3 years post-CABG
  Including death resulting from an acute myocardial infarction , sudden cardiac death, death due to heart failure, death due to stroke, death due to cardiovascular procedures, death due to cardiovascular hemorrhage, and death due to other cardiovascular causes
Myocardial infraction | 7 days, 30 days, 1 year, and 3 years post-CABG
  According to the 2017 Cardiovascular and Stroke Endpoint Definitions for Clinical Trials, including CABG-related MI, non CABG-related MI, silent MI and unknown type.
Stroke | 7 days, 30 days, 1 year, and 3 years post-CABG
  According to the 2017 Cardiovascular and Stroke Endpoint Definitions for Clinical Trials, including ischemic, hemorrhagic and unknown type.
Repeat revascularization | 7 days, 30 days, 1 year, and 3 years post-CABG
  According to the 2017 Cardiovascular and Stroke Endpoint Definitions for Clinical Trials, including any PCI and CABG.

CONTACTS AND LOCATIONS:
Overall Officials: Qiang Zhao, MD, Principal Investigator — Ruijin Hospital; Yunpeng Zhu, MD, Principal Investigator — Ruijin Hospital
Locations (1):
- Ruijin Hospital Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Xia T, Li B, Zhang W, Wang Z, Ye X, Zhou M, Li H, Qiu J, Zhu Y, Zhao Q. Risk factors for major adverse cardiovascular events after coronary artery bypass grafting using radial artery grafts. Front Cardiovasc Med. 2023 Sep 27;10:1238161. doi: 10.3389/fcvm.2023.1238161. eCollection 2023. PMID 37829689